CLINICAL TRIAL: NCT00430313
Title: Effects of Acupoint Electro-stimulation on Preventing Nausea and Vomiting Induced by Cisplatin or Oxaliplatin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0735; U19 CA12150301 (Other Grant/Funding Number: NCI); NCI-2012-02114 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Liver Cancer; Liver Metastasis
Keywords: Nausea; Vomiting; Electro-Stimulation; ES; K1 Acupuncture Point; Yongquan Acupuncture Point; TAI; transarterial infusion; liver metastasis; chemotherapy induced nausea and vomiting; CINV; Cisplatin; Oxaliplatin
MeSH Terms: conditions — Liver Neoplasms; Nausea; Vomiting | interventions — Acupuncture Points

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-Stimulation (Active Site) (Experimental): Electro-stimulation at an active (responsive) acupuncture site on the bottom of the foot.
  Interventions: Procedure: Electro-Stimulation of Yongquan (K1) Acupoint
- Electro-Stimulation (Inactive Site) (Experimental): Electro-stimulation at a inactive site on the bottom of the foot (a "placebo" site).
  Interventions: Procedure: Electro-Stimulation of Yongquan (K1) Acupoint

INTERVENTIONS:
Procedure: Electro-Stimulation of Yongquan (K1) Acupoint — Electro-stimulation at an active (responsive) acupuncture site on the bottom of the foot.
  Other Names: ES
  Arms: Electro-Stimulation (Active Site)
Procedure: Electro-Stimulation of Yongquan (K1) Acupoint — Electro-stimulation at a inactive site on the bottom of the foot (a "placebo" site).
  Other Names: ES
  Arms: Electro-Stimulation (Inactive Site)

SUMMARY:
Objectives:

This protocol is part of a larger grant funded by the NCI to create an international research center to study Traditional Chinese Medicine (TCM). All of the patients enrolled in this study will be treated at the Cancer Hospital, Fudan University, investigator's sister institution in Shanghai, China. No patients will be seen at MDACC. This protocol will be overseen by the Fudan University Institutional Review Board (IRB00002408) which has Federal Wide Assurance through the U.S. Department of Health & Human Services (Approved: April 25, 2002). The research nurses have received training at MDACC and will receive regular oversight by MDACC personnel.

The purpose of this randomized, placebo controlled study is to determine the effects of K1 acustimulation at controlling chemotherapy induced nausea and vomiting (CINV).

1. The primary aim of this study is to determine the effects of electro-stimulation of Yongquan (K1) acupoint on preventing nausea and vomiting induced by cisplatin or oxaliplatin.
2. The secondary aim is to observe the effects of electro-stimulation (ES) of Yongquan (K1) acupoint on pain, insomnia, abdominal distention, dizziness, and general sense of well-being.

DETAILED DESCRIPTION:
Nausea and vomiting are common side effects caused by chemotherapy. Some studies have shown that acupuncture can be helpful in treating nausea and vomiting. Acupuncture uses very thin needles inserted at certain points on the body that are believed to affect bodily functions. Researchers want to study the effects on nausea and vomiting of giving electro-stimulation (using wires attached to the body to provide very small electrical shocks to the skin) to an acupuncture site, compared to giving electro-stimulation to a inactive site (a site that does not respond to acupuncture).

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to be in 1 of 2 groups. Participants in one group will receive electro-stimulation at an active (responsive) acupuncture site on the bottom of the foot. Participants in the other group will receive electro-stimulation at a inactive site on the bottom of the foot (a "placebo" site).

Participants in both groups will have electro-stimulation on the feet. You will sit or lie down in bed. The acupuncturist will wet the points with a cotton ball dipped in water and attach the electrodes of the electro-stimulating instrument to the bottom of your feet. The electrodes are little paddles that will be attached with tape. The acupuncturist will begin slowly increasing the stimulation to a level you can withstand comfortably. This will last about 30 minutes.

The stimulation will occur about 1-2 hours before your TAI chemotherapy on the first day, and then between 7-9 A.M. on the next 5 days.

After each electro-stimulation procedure, your vital signs will be measured, you will complete quality-of-life questionnaires, and you will be asked about hiccups and diet tolerance (how nausea has affected your ability to eat or how much you eat). After your last electro-stimulation, you will also have a TCM diagnosis. This will include diagnosis by a doctor as well as by using a heart-rate machine and taking a photograph of your tongue. Blood (about 1 teaspoon) will also be drawn to check your liver function about 6 days after the treatments.

You will be given the standard medicines if you experience uncontrolled nausea or vomiting while on this study.

Your total participation on this study will last less than 2 weeks.

This is an investigational study. Up to 100 patients will take part in this study. All will be enrolled at the Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who will undergo TAI (transarterial infusion) for liver primary or other primary with liver metastasis
2. Between 18-75 years old
3. Patients who will receive TAI using cisplatin or oxaliplatin
4. Must give informed consent
5. If patients is female and of child bearing potential, must have a negative urine pregnancy test

Exclusion Criteria:

1. Has local skin infections at or near the acupoints
2. Previous TAI treatment using platinum-based chemotherapy
3. History of cerebrovascular or cardiovascular accident or spinal cord injury
4. Nausea and vomiting induced by intestinal obstruction
5. Has cardiac pacemaker
6. Mental incapacitation or significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry as these patients may not be able to cooperate with this slightly invasive procedure or with the data collection process
7. Currently using acupuncture
8. Vomiting or using 5-HT3 receptor antagonists or other antiemetic in 24 hours before TAI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01-04 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Level of Patient Nausea + Vomiting | 2 Years
  Vomiting and nausea will be classified according to the WHO criteria. The four levels of nausea are defined as: 0=no nausea, 1=slight nausea, 2=obvious nausea affecting normal life, and 3-4=continual and serious nausea. The four levels of vomiting are defined as: 0=no vomiting, 1=vomiting 1-2 times/day, 2=vomiting 2-4 times/day, and 3-4=vomiting 5 times/day.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org